CLINICAL TRIAL: NCT02282228
Title: Detecting Chronic Subdural Hematoma With Microwave Technology - An Open Study Evaluating the Sensitivity and Specificity of a Microwave-based Device, Medfield Strokefinder MD100, to Detect Chronic Subdural Hematoma
Brief Title: Detecting Chronic Subdural Hematoma With Microwave Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Medfield Diagnostics (Industry); Chalmers University of Technology (Other)
Responsible Party: Principal Investigator, Dr Thomas Skoglund, Principal Investigator, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CSH 01
Record Dates: First submitted 2014-10-22; First posted 2014-11-04 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Chronic Subdural Hematoma; Healthy Volunteers
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Medfield Strokefinder MD100 — Measurement with Medfield Strokefinder MD100.

SUMMARY:
An open study evaluating the sensitivity and specificity of a microwave-based device, Medfield Strokefinder MD100, to detect chronic subdural hematoma, by comparing measurements on patients recruited for surgery of chronic subdural hematoma to an age- and gender-matched group of healthy volunteers.

DETAILED DESCRIPTION:
This open study will enroll patients admitted for surgery of chronic subdural hematoma at the Department of Neurosurgery at Sahlgrenska University Hospital and compare them to measurements of healthy volunteers. Patients will be asked to participate in the study, as early as possible after admission. After physical examination, checking the inclusion/exclusion criteria, and after informed consent has been acquired, the microwave-based measurement will be performed. The diagnostic procedure is estimated to take 30 min whereof total subject measurement time will be less than five minutes. Healthy volunteers will be recruited in parallel and the same procedure as for the patients will be followed.

Safety will be followed throughout the study, and a safety follow-up will be performed 12 hours after the microwave-based investigation is finalized.

To avoid measurement bias all measurements, for both patients and healthy volunteers, will be performed by the same operator.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for surgery of chronic subdural hematoma.
* A CT scan of the patient has been performed, within the latest 96 hours.
* The patient should be able to have a normal conversation and understand the information about the study, corresponding to Glasgow Coma Scale (Verbal Response) of 5.
* Patient/healthy volunteer should be ≥ 18 years of age.
* The patient/healthy volunteer has signed a written informed consent.

Exclusion Criteria:

* Females who are pregnant or breast feeding women.
* Patient/healthy volunteer has a shunt or other foreign object implanted in the brain.
* Patient/healthy volunteer participating in any other clinical study that could interfere with the result in the ongoing study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for distinguishing chronic subdural hematoma patients from healthy volunteers using a classification algorithm. | The diagnostic procedure has an estimated duration of 30 minutes.
  The diagnostic ability of the device is calculated using a leave-one-out cross-validation method.

SECONDARY OUTCOMES:
Correlation between subdural hematoma volumes estimated by CT and by mathematical analysis of microwave data. | The diagnostic procedure has an estimated duration of 30 minutes.
  Pearson's linear correlation coefficient is calculated by comparing subdural hematoma volumes estimated by analysis of CT image and by a mathematical analysis of the microwave data.
Classification accuracy for estimating the position of the subdural hematoma through a mathematical analysis of the microwave data. | The diagnostic procedure has an estimated duration of 30 minutes.
  The ability of the device to estimate location of subdural hematoma is evaluated using a classification algorithm and leave-one-out cross validation.
Mean (± standard deviation) signal amplitude and phase shift caused by presence of chronic subdural hematoma. | The diagnostic procedure has an estimated duration of 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Skoglund, MD, PhD, Principal Investigator — Sahlgrenska University Hospital, Department of Neurosurgery
Locations (1):
- Sahlgrenska University Hospital, Department of Neurosurgery, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Result] Ljungqvist J, Candefjord S, Persson M, Jonsson L, Skoglund T, Elam M. Clinical Evaluation of a Microwave-Based Device for Detection of Traumatic Intracranial Hemorrhage. J Neurotrauma. 2017 Jul 1;34(13):2176-2182. doi: 10.1089/neu.2016.4869. Epub 2017 Mar 13. PMID 28287909